CLINICAL TRIAL: NCT00267215
Title: A One-week Multicenter, Multiple-dose, Randomized, Double-blind, Double-dummy, Parallel-group Comparison of the Analgesic Efficacy and Safety of Lumiracoxib (COX189), Celecoxib, and Placebo in the Treatment of Osteoarthritis of the Knee
Brief Title: Efficacy and Safety of Lumiracoxib
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCOX189A2301
Record Dates: First submitted 2005-12-16; First posted 2005-12-20 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-05

CONDITIONS: Osteoarthritis
Keywords: Lumiracoxib; osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — lumiracoxib

INTERVENTIONS:
Drug: Lumiracoxib

SUMMARY:
This trial assessed the safety and efficacy of a single dose of lumiracoxib 400 mg compared to placebo and to a single dose of celecoxib 200mg. It also assessed safety and efficacy of 400mg lumiracoxib administered once a day for 7 days compared to placebo and to 200 mg celecoxib twice daily.

ELIGIBILITY:
Inclusion criteria:

* Osteoarthritis of the knee
* Pain intensity at baseline of at least 50mm on a 100mm visual analog scale

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 330
Dates: Start 2000-11; Primary Completion 2001-02 (Actual)

PRIMARY OUTCOMES:
Assess the short-term (3-5 hours) analgesic efficacy of COX189, 400mg administered once a day for 7 days, compared to placebo and to 200mg celecoxib bid

SECONDARY OUTCOMES:
Assess the safety and tolerability profile of COX189 in comparison to placebo and celecoxib

CONTACTS AND LOCATIONS:
Locations (1):
- Novartis, Nuremberg, Germany

REFERENCES:
- [Derived] Wittenberg RH, Schell E, Krehan G, Maeumbaed R, Runge H, Schluter P, Fashola TO, Thurston HJ, Burger KJ, Trechsel U. First-dose analgesic effect of the cyclo-oxygenase-2 selective inhibitor lumiracoxib in osteoarthritis of the knee: a randomized, double-blind, placebo-controlled comparison with celecoxib [NCT00267215]. Arthritis Res Ther. 2006;8(2):R35. doi: 10.1186/ar1854. Epub 2006 Jan 16. PMID 16469112